CLINICAL TRIAL: NCT06124534
Title: Bilateral Occipital Nerve Field Stimulation for the Prophylactic Treatment of Difficult-to-treat Chronic Cluster Headache
Brief Title: Bilateral Occipital Nerve Field Stimulation for the Treatment of dtCCH
Acronym: BONS
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: device upgrade/requires competent authority approval
Sponsor: Man and Science, SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOC-130
Record Dates: First submitted 2023-10-26; First posted 2023-11-09 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Chronic Cluster Headache
Keywords: Cluster Headaches
MeSH Terms: conditions — Cluster Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blistim System (Experimental): Occipital Nerve Stimulation using the BliStim Occipital Nerve Stimulator
  Interventions: Device: Neurostimulation of the Occipital Nerve Field

INTERVENTIONS:
Device: Neurostimulation of the Occipital Nerve Field — BliStim Neurostimulation system

SUMMARY:
The purpose of this study is to assess the initial safety, tolerability, and effectiveness of the novel BliStim occipital nerve field stimulation therapy for the prevention of chronic cluster headaches. This is a prospective, first in human study.

ELIGIBILITY:
Inclusion Criteria:

1. ICHD-3 criteria for chronic cluster headache
2. Documented history of CCH since at least 2 years
3. Minimum mean attack frequency of 4 attacks per week
4. Age range: 18-70 years
5. Difficult-to-treat CCH with documented previous complete failure, insufficient efficacy, intolerance, or contra-indications to most preventive CH treatments among which are oral steroids or suboccipital infiltrations, verapamil, lithium carbonate and topiramate.
6. No preventive CH treatment or stable preventive CH medication for ≥ 2 weeks before enrolment. Subject agrees not to change existing treatment during the whole duration of the trial.
7. Subject written informed consent provided before enrolment
8. Subject willing and capable of subjective evaluation and to fill in an electronic CH diary, to understand questionnaires, and to read, understand and sign the written informed consent form.
9. Subject willing and able to comply with study-related requirements, procedures, and visits.

Exclusion Criteria:

1. Other significant neurological, psychiatric, or disabling diseases which in the opinion of the investigator may interfere with the study.
2. History of epilepsy, current treatment of epilepsy
3. Documented history of cerebrovascular accident (CVA)
4. Subjects suffering from a substance use disorder, as defined by Diagnostic and Statistical Manual of Mental Disorders (DSM) criteria. Recreational use of cannabis is allowed.
5. Subjects at high risk of suicide/suicidal ideation in the past one year assessed with the C-SSRS
6. Having another active implanted device such as a cardiac pacemaker, a spinal cord, peripheral nerve, sphenopalatine ganglion, or deep brain hypothalamic stimulator, and/or a drug delivery pump, etc.
7. Cranial botulinum toxin injections in the past 3 months before enrolment. Administration of the following treatments in the last month before enrolment: monoclonal antibodies blocking calcitonin gene-related peptide transmission, suboccipital infiltrations with steroids and/or local anaesthetics, oral steroids, radiofrequency procedure or infiltrations of the sphenopalatine ganglion, opioids WHO 3.
8. Medication overuse headache (ICHD 3 8.2)
9. Inability to fill out an electronic diary.
10. Previous surgery or trauma involving the cervical spine or the occipital bone
11. Coagulopathy or required anticoagulant medications that cannot be safely discontinued in the perioperative period.
12. Concurrent participation in another clinical study
13. Planned pregnancy, pregnancy, or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2024-11-21 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Safety Evaluation of the Device [Time Frame:12 weeks / 48 weeks] | 12-weeks post implantation and through study completion at 48 weeks
  The primary endpoint is safety and is assessed through the incidence of procedure related and/or device-related adverse events during the 12-weeks post implantation and the rate of all adverse events during the entire 48-week study period.

CONTACTS AND LOCATIONS:
Overall Officials: J-P Van Buyten, Principal Investigator — VITAZ Hospital, Sint Niklaas, Belgium
Locations (1):
- VITAZ Hospital, Sint-Niklaas, Belgium

IPD SHARING:
Plan to Share IPD: No